CLINICAL TRIAL: NCT06072404
Title: Comparative Analysis of Different Protocols for Dental Exactions in Patients at Risk of MRONJ: Case-control Study
Brief Title: OZONE_EXO: Comparative Analysis of Protocols for Dental Exactions in Patients at Risk of MRONJ: Case-control Study
Acronym: OZONE_EXO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Olga Di Fede, Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OZONE_EXO
Record Dates: First submitted 2023-09-27; First posted 2023-10-10 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: MEDICATION RELATED OSTEONECROSIS OF THE JAW
Keywords: MRONJ; Osteonecrosis; Ozone therapy; Jaw; Antiresorptive; Antiangiogenic drugs; Adverse event
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (OZONE_EXO) (Experimental): intra-tissutal perialveolar injections of a 15-mL mixture of OxigenOzone (O2O3) with a 26Gx1⁄2 - 0.45x13 mm needle and insufflation of the same mixture in the post-extraction site in patients at risk of medication-induced osteonecrosis of the jaw (ONJ).
  Interventions: Biological: OxigenOzone_Insufflation
- Group B (NO_OZONE_EXO) (No Intervention): Tooth extraction in patients at risk of medication-induced osteonecrosis of the jaw (ONJ) without the use of ozone application.

INTERVENTIONS:
Biological: OxigenOzone_Insufflation — intra-tissutal perialveolar injections of a 15-mL mixture of OxigenOzone (O2O3) with a 26Gx 1⁄2 - 0.45x13 mm needle and insufflation of the same mixture in the post-extraction site for at least 1 minute, hemostasis, and suture.
  Arms: Group A (OZONE_EXO)

SUMMARY:
Medication-related osteonecrosis of the jaw (MRONJ) is a serious adverse reaction of antiresorptive and antiangiogenic agents; it is also a potentially painful and debilitating condition. Today, no specific studies have prospectively evaluated the efficacy of its treatment and no robust standard of care has been established.

Among non-invasive procedures to treat MRONJ, the use of medical ozone (O3) arises for its properties and has been deployed and evaluated. O3 has generally proven to play a role in the treatment of chronic, nonhealing, or ischemic wounds, due to its antimicrobial and anti-oxidant properties and to bio-stimulation; it has been extensively used for different medical approaches and purposes. In oral cavity, local applications are carried out by ozonized water (i.e. spray or compress) or gel.

The aim of this study was to carry out a case-control study in order to compare two different protocols of dental extractions in patients at risk of MRONJ, with and without infiltration of a mixture of oxygen-ozone.

All the cases in our study are cancer and oncologic and osteometabolic patients undergoing high-risk therapy for MRONJ (antiresorptive and antiangiogenic drugs) who require dental extractions with a poor prognosis. During the first examination (T0), medical, pharmacological, and dental history of patients are recorded. Data collected are: (1) age; (2) gender; (3) indications for use, type, cumulative dose and duration of MRONJ-related drugs; (4); history of chemotherapy; (5) other medications; (6) other diseases; (7) smoking.

For each patient, an orthopantomography and a cone beam computed tomography of the teeth are performed only if indicated.

DETAILED DESCRIPTION:
The enrolled patients were randomly divided into two groups:

Group A: consisting of 38 patients (undergoing ozone treatment) (OZONE_EXO) intra-tissutal perialveolar injections of a 15-mL mixture of OxigenOzone (O2O3) with a 26Gx1⁄2 - 0.45x13 mm needle and insufflation of the same mixture in the post-extraction site in patients at risk of medication-induced osteonecrosis of the jaw (ONJ).

Group B: comprising 79 controls (not undergoing ozone treatment).(NO_OZONE_EXO) Tooth extraction in patients at risk of medication-induced osteonecrosis of the jaw (ONJ) without the use of ozone application.

Following the same approach as in Group A, patients in Group B underwent additional follow-up visits at T1 (3-5 days), T2 (14 days), and T3 (6 weeks) post-extraction, in accordance with Inflammatory - P roliferative - Remodeling (IPR) Wound Healing Scale.

the IPR scale score, to meticulously monitor surgical wound healing and record pain intensity using the NRS scale, rather than the originally planned VAS scale, for enhanced ease of use [22].

The IPR scale provided a comprehensive assessment of wound healing through distinct subscales, each ranging from 0 to 1, resulting in a total score ranging from 0 to 16. These subscales evaluated the inflammatory response, proliferative response, and remodeling process. At the conclusion of the follow-up period, the total IPR score was computed, with scores spanning from 0 to 16. Scores of 0-4 denoted poor healings, scores of 5-10 indicated acceptable healing, while scores of 11-16 suggested excellent healing.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 yrs
* patients at risk of developing MRONJ for previous or current administration of drugs related
* extraction of teeth with a poor prognosis due to severe decay and/or periodontitis

Exclusion Criteria:

* previous radiation in the head and neck area
* neoplastic involvement of the jaw
* previous MRONJ diagnosis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Di Fede, Professor, Principal Investigator — University of Palermo
Locations (1):
- Azienda Ospedaliera Universitaria Policlinico "P. Giaccone" Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campisi G, Mauceri R, Bertoldo F, Bettini G, Biasotto M, Colella G, Consolo U, Di Fede O, Favia G, Fusco V, Gabriele M, Lo Casto A, Lo Muzio L, Marciano A, Mascitti M, Meleti M, Mignogna MD, Oteri G, Panzarella V, Romeo U, Santarelli A, Vescovi P, Marchetti C, Bedogni A. Medication-Related Osteonecrosis of Jaws (MRONJ) Prevention and Diagnosis: Italian Consensus Update 2020. Int J Environ Res Public Health. 2020 Aug 18;17(16):5998. doi: 10.3390/ijerph17165998. PMID 32824826
- [Background] Oldoini G, Frabattista GR, Saragoni M, Cosola S, Giammarinaro E, Genovesi AM, Marconcini S. Ozone Therapy for Oral Palatal Ulcer in a Leukaemic Patient. Eur J Case Rep Intern Med. 2020 Jan 14;7(2):001406. doi: 10.12890/2020_001406. eCollection 2020. PMID 32133312
- [Background] Palma LF, Joia C, Chambrone L. Effects of ozone therapy on periodontal and peri-implant surgical wound healing: a systematic review. Quintessence Int. 2023 Feb 10;54(2):100-110. doi: 10.3290/j.qi.b3512007. PMID 36437805
- [Background] Agrillo A, Ungari C, Filiaci F, Priore P, Iannetti G. Ozone therapy in the treatment of avascular bisphosphonate-related jaw osteonecrosis. J Craniofac Surg. 2007 Sep;18(5):1071-5. doi: 10.1097/scs.0b013e31857261f. PMID 17912085

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were identified among patients attending the "Oral Medicine with Dentistry for Fragile Patients Unit" at the Paolo Giaccone Policlinico University Hospital of Palermo from February 2018 to March 2020. Patients were approached with written and verbal information about the study.
Pre-assignment Details: The study recruited 117 patients (27 male and 90 female) and were randomized to treatment.
Period: Overall Study
Arm/Group | Group A (OZONE_EXO) | Group B (NO_OZONE_EXO)
Started | 38 | 79
Completed | 38 | 79
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (OZONE_EXO) | Group B (NO_OZONE_EXO) | Total
Number analyzed (Participants) | 38 | 79 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 79 | 117
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 63 | 90
  Male | 11 | 16 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 79 | 117
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 38 | 79 | 117

OUTCOME MEASURES:

1. Primary Outcome: Healing Evaluation Using Inflammatory-Proliferative-Remodelling Scale (IPR Scale): Inflammatory Phase
Description: The inflammatory phase is evaluated 3-5 days after tissue injury on the basis of eight parameters, measured on a 9-point scale (0-8): bleeding (spontaneously or on palpation), granulation tissue, hematoma, tissue color, incision margins, suppuration, edema, and pain. A score of 5-8 indicates a successful inflammatory phase
Time Frame: 3-5 days after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A (OZONE_EXO) | Group B (NO_OZONE_EXO)
Number analyzed (Participants) | 38 | 79
score on a scale | 2 (0.87) | 2.49 (0.875)

2. Primary Outcome: Healing Evaluation Using Inflammatory-Proliferative-Remodelling Scale (IPR Scale): Proliferative Phase:
Description: The proliferative phase is evaluated 14 days after tissue injury on the basis of five parameters, measured on a 6-point scale (0-5): re-epithelialization, tissue color, scar, suppuration, and pain. A score of 3-5 score indicates successful healing.
Time Frame: 14 days after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A (OZONE_EXO) | Group B (NO_OZONE_EXO)
Number analyzed (Participants) | 38 | 79
score on a scale | 4.24 (1.51) | 3.7 (1.02)

3. Primary Outcome: Healing Evaluation Using Inflammatory-Proliferative-Remodelling Scale (IPR Scale): Remodelling Phase
Description: The remodeling phase is evaluated 6 weeks after tissue injury on the basis of three parameters, measured on a 4-point scale (0-3): scar, tissue color, and pain. A score of 2-3 indicates successful healing
Time Frame: 6 weeks after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A (OZONE_EXO) | Group B (NO_OZONE_EXO)
Number analyzed (Participants) | 38 | 79
score on a scale | 3 (0) | 2.96 (0.192)

4. Secondary Outcome: Healing Evaluation Using IPR Scale: Total Process
Description: The total score of the IPR scale ranges from 0 to 16:0-4 indicates poor healing; 5-10, acceptable healing; and 11-16, excellent healing The inflammatory phase carries the greatest weight in the final score because its impairment can jeopardize the entire series of biologic events leading to early wound healing.
Time Frame: 6 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A (OZONE_EXO) | Group B (NO_OZONE_EXO)
Number analyzed (Participants) | 38 | 79
score on a scale | 9.37 (1.79) | 9.15 (1.38)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Group A (OZONE_EXO) | Group B (NO_OZONE_EXO)
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/79
Other Adverse Events (participants affected / at risk) | 0/38 | 0/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (OZONE_EXO) (N=38) | Group B (NO_OZONE_EXO) (N=79)
Osteonecrosis of the jaw (Infections and infestations) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT06072404/Prot_SAP_000.pdf